CLINICAL TRIAL: NCT04624932
Title: Early Childhood Outside (ECO) Early Childhood Educator (ECE) Tool - Randomized Controlled Trial Study
Brief Title: Early Childhood Outside (ECO) - Randomized Controlled Trial Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Lawson Foundation (Other)
Responsible Party: Principal Investigator, Mariana Brussoni, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H19-03644
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Risk Assessment; Online Intervention; Child Development
Keywords: Risk reframing tool; Children's outdoor play; Children's outdoor risky play; Early childhood education

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocations will be concealed to the researchers at participant assignment and data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk Reframing (RR) Digital Tool (Experimental): Participants proceed through three chapters in the tool: https://outsideplay.ca.
  Chapter 1: reflecting on their own childhood play activities; what they got out of these experiences; outdoor play activities of the children at their center; what they do to promote children's outdoor play; what gets in the way in promoting children outdoor play.
  Chapter 2: imagining themselves in six video segments where they must decide how to communicate with parents; and, whether they allow children to engage in rough and tumble play, play at heights, play with tools, play at speed/mud play, and resolve conflicts amongst themselves
  Chapter 3: reflecting on their barriers and things that helped them promote and support the children's outdoor play at their center. Participants to assess whether there is anything they want to change to set a realistic goal, outlining steps for attaining that goal.
  Interventions: Behavioral: RR Digital Tool
- Position Statement on Active Outdoor Play (Sham Comparator): The position statement summarizes the issues and research regarding children's access to outdoor play and provides recommendations for various stakeholders. It states that "access to active play in nature and outdoors - with its risks - is essential for healthy child development" and recommends increasing children's opportunities for self-directed play in all settings. The Position Statement includes recommendations for parents, educators, health professionals, administrators and various level of governments to address the barriers to children's outdoor play.
  It addresses common misconceptions and encourages that danger be differentiated from risk and outdoor play and fun be valued as much as safety.
  Interventions: Behavioral: Position Statement on Active Outdoor Play

INTERVENTIONS:
Behavioral: RR Digital Tool — This is the intervention condition. Participants in this condition will take the RR digital tool available at https://outsideplay.ca.
  Arms: Risk Reframing (RR) Digital Tool
Behavioral: Position Statement on Active Outdoor Play — This is the control condition. Participants in this condition will read the position statement that summarizes the issues and research regarding children's access to outdoor play.
  Arms: Position Statement on Active Outdoor Play

SUMMARY:
Outdoor play is important for children as it can promote healthy social and physical development, emotional well-being, self-confidence, risk management and overall physical activity. Yet, opportunities for outdoor play have been decreasing across generations due to perceptions that it is dangerous and unnecessary. Early childhood educators (ECEs) and administrators are struggling to provide children with high quality and stimulating outdoor play time. To help ECEs and administrators, the investigators have developed a Risk Reframing (RR) digital tool, https://outsideplay.ca, which is underpinned by social cognitive theory (SCT) and health behaviour change techniques.

The aim of the current study is to test the efficacy of the RR digital tool in: 1) increasing ECEs/administrators' tolerance of risk in play; and, 2) attaining their behavior change goal in promoting children's outdoor play at their early childcare center.

The investigators will conduct a single-blind (researchers and outcome assessors) randomized controlled trial and will obtain complete data on at least 206 early childhood educators and administrators currently working in Canada. The RR digital tool is designed for a one-time visit and includes three chapters of self-reflection and experiential learning tasks. The control condition consists of reading the Position Statement on Active Outdoor Play, a 2-page information sheet on children's active outdoor play.

Primary outcome is increased tolerance of risk in play, as measured by the Tolerance of Risk in Play Scale - teacher version. Secondary outcome is self-reported attainment of a behaviour change goal that participants set for themselves. The investigators will test the hypothesis that there will be differences between the intervention and control conditions with respect to tolerance of risk in play and goal attainment.

DETAILED DESCRIPTION:
The study uses 2-condition (control and intervention) randomized controlled trial design.

Participants will be recruited through advertising on social media, distributing notices throughout networks, and snowball sampling. The aim is to obtain complete data on 206 participants, thus the investigators will try to recruit at least 324 ECEs and administrators at baseline to account for attrition. The investigators considered 75% and 85% retention rate at 1-week post-intervention and 3-months post-intervention, respectively. Interested participants will complete a questionnaire in REDCap electronic data capture tool hosted at British Columbia Children's Hospital Research Institute to answer eligibility questions and provide informed consent. Enrolled participants will be sent a link to the baseline questionnaire package to be completed in REDcap. Demographic questions are asked to understand the general background of participants (e.g., sex, age) and their ECE center (e.g., approximately how many staff are at their center).

They will then be randomly assigned to one of the two conditions: 1) Control condition, or, 2) Intervention condition. Neither the researchers nor participants will know in advance which condition participants will be assigned to. There is a 50% chance that they are assigned to either condition. The randomization schedule will be generated beforehand in sealedenvelop.com using blocks of size 2, 4, 6. The list will be then transferred to REDCap. Participants will not be blinded to allocation, because the nature of the intervention does not allow it. Allocation will be concealed to the researchers at participant assignment as well as data analysis.

Participants who are assigned to Control condition will be provided with a PDF version of the position statement on active outdoor play, which can take up 20 minutes to read. Then, they will be invited to set a goal that could help them give children at their center more opportunities for outdoor play.

Participants who are assigned to Intervention condition will be automatically taken to the online tool, https://outsideplay.ca. The online tool is to reframe participants' perceptions of outdoor play and change their service delivery. It includes a series of interactive video scenarios where participants can make choices, which will result in different endings for each scenario. This can take up to 100 minutes to complete. Then participants will be invited to set a goal that could help them give children at their center more opportunities for outdoor play.

Participants who are assigned to Control condition will have access to the online tool upon completion of their participation in the current study.

After 1-week, all participants who completed the baseline survey and the intervention (e.g., the Position Statement on Active Outdoor Play or the RR tool) will receive an email inviting them to complete a follow-up survey questionnaire. The investigators will also follow up on whether they had accomplished their goal.

After 3-months, all participants who completed the 1-week post-intervention survey will receive another email to complete the same follow-up survey questionnaire for the final time. The investigators will also follow up on whether they had accomplished their goal.

The study hypotheses are:

1. Participants in Intervention condition will have a significantly greater increase of tolerance for risk in play than participants in Control condition.
2. A greater proportion of participants in Intervention condition will attain their behavior change goal, than participants in Control condition.

ELIGIBILITY:
Inclusion Criteria:

1. Being 19 years of age or older;
2. Currently working or training in the early childhood education field in Canada; and,
3. Being able to speak, read, and understand English.
4. Having access to the internet

Exclusion Criteria:

n/a

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 563 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Brussoni, Principal Investigator — University of British Columbia / BC Children's Hospital
Locations (1):
- British Columbia Children's Hospital Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The data set will be available from Dr. Brussoni upon reasonable requests.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting upon publication of the RCT results until five years after publication.
Access Criteria: Dr. Brussoni will review requests and share supporting information as indicated above with researchers and students going similar research.

REFERENCES:
- [Background] Tremblay MS, Gray C, Babcock S, Barnes J, Bradstreet CC, Carr D, Chabot G, Choquette L, Chorney D, Collyer C, Herrington S, Janson K, Janssen I, Larouche R, Pickett W, Power M, Sandseter EB, Simon B, Brussoni M. Position Statement on Active Outdoor Play. Int J Environ Res Public Health. 2015 Jun 8;12(6):6475-505. doi: 10.3390/ijerph120606475. PMID 26062040
- [Background] ParticipACTION. The Biggest Risk Is Keeping Kids Indoors: ParticipACTION Report Card on Physical Activity for Children and Youth. Toronto, Ontario; 2015
- [Background] Ihrig KM. Teacher tolerance of risk in play scale (T-TRiPS): Evaluating the psychometric properties of a new measure. (Unpublished master thesis). Colorado State University, Fort Collins, Colorado, USA; 2020.
- [Derived] Brussoni M, Han CS, Lin Y, Jacob J, Munday F, Zeni M, Walters M, Oberle E. Evaluation of the Web-Based OutsidePlay-ECE Intervention to Influence Early Childhood Educators' Attitudes and Supportive Behaviors Toward Outdoor Play: Randomized Controlled Trial. J Med Internet Res. 2022 Jun 10;24(6):e36826. doi: 10.2196/36826. PMID 35687394
- [Derived] Brussoni M, Han CS, Jacob J, Munday F, Zeni M, Walters M, Cheng T, Schneeberg A, Fox E, Oberle E. A Web-Based Risk-Reframing Intervention to Influence Early Childhood Educators' Attitudes and Supportive Behaviors Toward Outdoor Play: Protocol for the OutsidePlay Study Randomized Controlled Trial. JMIR Res Protoc. 2021 Nov 18;10(11):e31041. doi: 10.2196/31041. PMID 34792479

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants between December 1, 2020 to March 15, 2021 via social media posts - FaceBook, FaceBook Ads, Twitter and Instagram - and mass email through partner and professional networks.
Pre-assignment Details: Eligible participants provided consent by downloading the consent form and selecting a checkbox to participate. Enrolled participants completed the baseline survey (demographic, and, a questionnaire on tolerance for risk in play, self-efficacy, and stage of change) and entered their email addresses. Then, we automatically randomized enrolled participants in the REDCap to one of the two conditions: intervention and control. Participants had an equal likelihood of being assigned to each condition.
Groups:
- Position Statement on Active Outdoor Play: Position Statement Active Outdoor Play: The position statement summarizes the issues and research regarding children's access to outdoor play and provides recommendations for various stakeholders. It states that "access to active play in nature and outdoors - with its risks - is essential for healthy child development" and recommends increasing children's opportunities for self-directed play in all settings. The Position Statement includes recommendations for parents, educators, health professionals, administrators and various level of governments to address the barriers to children's outdoor play. It addresses common misconceptions and encourages that danger be differentiated from risk and outdoor play and fun be valued as much as safety.
- Risk Reframing (RR) Digital Tool: RR Digital Tool: This is the intervention condition. Participants in this condition completed the RR digital tool available at https://outsideplay.ca.
  Chapter 1: reflecting on their own childhood play activities; what they got out of these experiences; outdoor play activities of the children at their center; what they do to promote children's outdoor play; what gets in the way in promoting children outdoor play.
  Chapter 2: imagining themselves in six video segments where they must decide how to communicate with parents; and, whether they allow children to engage in rough and tumble play, play at heights, play with tools, play at speed/mud play, and resolve conflicts amongst themselves Chapter 3: reflecting on their barriers and things that helped them promote and support the children's outdoor play at their center. Participants to assess whether there is anything they want to change to set a realistic goal, outlining steps for attaining that goal.
Period: Overall Study
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool
Started | 282 | 281
1-week Post-intervention | 209 | 126
Completed | 195 | 119
Not Completed | 87 | 162

BASELINE CHARACTERISTICS:
Groups:
- Position Statement on Active Outdoor Play: Position Statement Active Outdoor Play: The position statement summarizes the issues and research regarding children's access to outdoor play and provides recommendations for various stakeholders. It states that "access to active play in nature and outdoors - with its risks - is essential for healthy child development" and recommends increasing children's opportunities for self-directed play in all settings. The Position Statement includes recommendations for parents, educators, health professionals, administrators and various level of governments to address the barriers to children's outdoor play. It addresses common misconceptions and encourages that danger be differentiated from risk and outdoor play and fun be valued as much as safety (ParticipACTION Canada, 2015; Tremblay et al., 2015).
- Total: Total of all reporting groups
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool | Total
Number analyzed (Participants) | 282 | 281 | 563
Age, Customized [Count of Participants; unit: Participants]
  19-24 years | 26 | 33 | 59
  25-30 years | 72 | 55 | 127
  31-40 years | 71 | 86 | 157
  41-50 years | 66 | 64 | 130
  51 years and older | 46 | 42 | 88
  Participant did not provide answer | 1 | 1 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 272 | 272 | 544
  Non-female | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Canada: British Columbia | 129 | 129 | 258
  Canada: New Brunswick | 52 | 44 | 96
  Canada: Ontario | 64 | 66 | 130
  Canada: Others | 36 | 40 | 76
  Canada: Participant did not provide answer | 1 | 2 | 3
Language [Count of Participants; unit: Participants]
  English | 263 | 261 | 524
  Others | 19 | 20 | 39
Role [Count of Participants; unit: Participants]
  Early childhood educator (ECE) | 203 | 189 | 392
  ECE administrator | 75 | 90 | 165
  Others | 4 | 2 | 6
Years working in the field [Mean (Standard Deviation); unit: years] | 10.22 (9.51) | 10.05 (9.16) | 10.14 (9.33)
Years working at the current center [Mean (Standard Deviation); unit: years] | 6.09 (7.41) | 5.18 (5.98) | 5.63 (6.74)
Whether the center is licensed [Count of Participants; unit: Participants]
  Yes | 266 | 264 | 530
  No | 7 | 7 | 14
  Participant did not provide answer | 9 | 10 | 19
Number of children at the center [Count of Participants; unit: Participants]
  Small: 1-24 | 91 | 95 | 186
  Medium: 25-48 | 76 | 78 | 154
  Large: >= 49 | 111 | 106 | 217
  Participant did not provide answer | 4 | 2 | 6
Number of staffs at the center [Count of Participants; unit: Participants]
  Small: 1-5 | 100 | 102 | 202
  Medium: 6-12 | 85 | 91 | 176
  Large: >= 13 | 91 | 82 | 173
  Participant did not provide answer | 6 | 6 | 12
Whether the center has a designated outdoor space for children [Count of Participants; unit: Participants]
  Yes | 270 | 270 | 540
  No | 8 | 9 | 17
  Participant did not provide answer | 4 | 2 | 6
Quality of the center's outdoor space for children [Count of Participants; unit: Participants]
  Very good | 96 | 88 | 184
  Good | 95 | 110 | 205
  Acceptable | 65 | 60 | 125
  Poor | 12 | 11 | 23
  Very poor | 2 | 0 | 2
  Participant did not provide answer | 12 | 12 | 24
Hours children spent playing outdoors at the center [Mean (Standard Deviation); unit: hours] | 2.01 (1.15) | 2.14 (1.13) | 2.08 (1.14)
Feeling supported by colleagues in general [Count of Participants; unit: Participants]
  Yes | 251 | 250 | 501
  No or others | 31 | 27 | 58
  Participant did not provide answer | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Tolerance of Risk in Play Across Baseline, 1-week Post-intervention and 3-months Post-intervention
Description: This scale measures participants' tolerance of risk in outside play. Teacher Tolerance of Risk in Play Scale has 26 items of yes/no (coded as 1 and 0, respectively) survey questions of risk tolerance. To account for item difficulty and respondent trait, we convert respondents' responses to a psychometric measure that is standardized to z-scores. We standardized the measure to z-scores at each measurement time point. For example, at baseline, all respondents' (including those from control and intervention group) psychometric measures have a population mean of zero/0 and standard deviation of 1. A higher z-score means a higher tolerance of risk in play (in the case of our study, a higher score means a more favorable outcome). In this table, we present the outcome measures as absolute z-score values, rather than change from two time points. We do not consider clinically relevant threshold for this outcome measure as there is no established literature.
Time Frame: Baseline, 1-week post-intervention, and 3-months post-intervention
Population: A total of 563 participants with baseline demographic and other survey data completed was included at baseline. Of 563 participants, 282 were randomized to the control group and 281 to the intervention group. At 1-week post-intervention, 335 participants were included; and at 3-month post-intervention, 314 participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool
Number analyzed (Participants) | 282 | 281
score on a scale
  Baseline outcome | 0.040 (1.207) | -0.040 (1.243)
  1-week post-intervention: number analyzed (Participants) | 209 | 126
  1-week post-intervention | -0.156 (1.304) | 0.262 (1.117)
  3-month post-intervention: number analyzed (Participants) | 195 | 119
  3-month post-intervention | -0.118 (1.400) | 0.200 (1.211)

2. Secondary Outcome: Change in Attainment of a Behavior Change Goal
Description: This is a yes/no self-report question asking participants if they think they had attained their behavior change goal. Unit of measure is 'yes' or 'no' to measure incidence of behavior change goal attainment.For the purpose of our analyses the category of "Yes" is an indication of behaviour change while the category of "No" is an indication of no behaviour change.
Time Frame: 1-week post-intervention, and 3-months post-intervention
Population: We included 335 participants with complete secondary outcome data (goal) at 1-week post-intervention, and 314 participants at 3-month post-intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool
Number analyzed (Participants) | 209 | 126
Participants
  1-week post-intervention: Yes | 141 | 94
  1-week post-intervention: No | 68 | 32
  3-months post-intervention: number analyzed (Participants) | 195 | 119
  3-months post-intervention: Yes | 163 | 106
  3-months post-intervention: No | 32 | 13

ADVERSE EVENTS:
Description: Adverse events were not monitored/assessed because this RCT was not clinical-based. It was to test the efficacy of a web-based intervention to change participants' perception of risk in children's outdoor play.
Arm/Group | Position Statement on Active Outdoor Play | Risk Reframing (RR) Digital Tool
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Given the nature of the interventions, it was not possible to blind participants to their allocation, thus potentially introducing sources of bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04624932/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT04624932/ICF_001.pdf